CLINICAL TRIAL: NCT03776175
Title: A PHASE 2A, RANDOMIZED, DOUBLE BLIND (SPONSOR-OPEN), PLACEBO CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE PHARMACODYNAMICS, SAFETY AND TOLERABILITY OF PF-05221304 AND PF-06865571 CO-ADMINISTERED FOR 6 WEEKS IN ADULTS WITH NON-ALCOHOLIC FATTY LIVER DISEASE (NAFLD)
Brief Title: A Study To Assess Pharmacodynamics, Safety And Tolerability Of PF-05221304 And PF-06865571 Co-Administered For 6 Weeks In Adults With Non-Alcoholic Fatty Liver Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C3711001
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (PF 05221304) BID Placebo (PF 06865571) BID
  Interventions: Drug: Placebo
- PF-05221304 Monotherapy (Experimental): 15 mg PF-05221304 BID Placebo (PF-06865571) BID
  Interventions: Drug: PF-05221304 Monotherapy; Drug: Placebo
- PF-06865571 Monotherapy (Experimental): Placebo (PF-05221304) BID 300 mg PF-06865571 BID
  Interventions: Drug: PF-06865571 Monotherapy; Drug: Placebo
- PF-05221304 and PF-06865571 Combination (Experimental): 15 mg PF-05221304 BID 300 mg PF-06865571 BID
  Interventions: Drug: PF-05221304 Monotherapy; Drug: PF-06865571 Monotherapy; Drug: PF-05221304 and PF-06865571 Combination

INTERVENTIONS:
Drug: PF-05221304 Monotherapy — Participants enrolled in this Arm will receive 15 mg dose of PF-05221304 (3 tablets of 5 mg each) and 3 tablets of Placebo for PF-06865571, each to be taken twice daily for 41 days and once on Day 42.
  Other Names: Arm B
  Arms: PF-05221304 Monotherapy; PF-05221304 and PF-06865571 Combination
Drug: PF-06865571 Monotherapy — Participants enrolled in this Arm will receive 300 mg dose of PF-06865571 (3 tablets of 100 mg each) and 3 tablets of Placebo for PF-05221304, all to be taken twice daily for 41 days and once on Day 42.
  Other Names: Arm C
  Arms: PF-05221304 and PF-06865571 Combination; PF-06865571 Monotherapy
Drug: Placebo — Participants enrolled in this Arm will receive 3 tablets for Placebo of PF-05221304 and 3 tablets of Placebo of PF-06865571, to be taken twice daily for 41 days and once on Day 42.
  Other Names: Arm A
  Arms: PF-05221304 Monotherapy; PF-06865571 Monotherapy; Placebo
Drug: PF-05221304 and PF-06865571 Combination — Participants enrolled in this Arm will receive 15 mg dose of PF-05221304 (3 tablets of 5 mg each) and 3 tablets of PF-06865571 (3 tablets of 100 mg each), each to be taken twice daily for 41 days and once on Day 42.
  Other Names: Arm D
  Arms: PF-05221304 and PF-06865571 Combination

SUMMARY:
This study is to assess the effect of PF 05221304 alone, PF 06865571 alone, the co administration of PF 05221304 and PF 06865571, or placebo on whole liver fat in subjects with NAFLD. In addition, this study will evaluate the safety and tolerability of co administration of PF 05221304 and PF 06865571 along with the effects on selected pharmacodynamics (PD)/exploratory parameters, compared to administration of PF 05221304 alone, PF 06865571 alone, and placebo in adults with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or female subjects of non childbearing potential
* Total body weight of >50 kg (110 lbs) and a BMI greater than or equal to 25 kg/m2
* Medical diagnosis of Type 2 Diabetes Mellitus (T2DM) being treated with no more than 1 acceptable oral antidiabetic drug OR Subjects without a diagnosis of T2DM that meet 2 or more of the following 5 criteria commonly associated with metabolic syndrome

  * Fasting Plasma Glucose (FPG) greater than or equal to 100 mg/dL;
  * Documentation of at least stage 1 hypertension or medical history of hypertension;
  * Fasting serum HDL C <40 mg/dL for males and <50 mg/dL for females, or on pharmacological agents with explicit purpose to increase HDL-C;
  * Fasting serum triglyceride (TG) greater than or equal to 150 mg/dL or on pharmacological agents with explicit purpose to decrease TG;
  * Waist circumference greater than or equal to 40 inches (102 cm) for males and 35 inches (89 cm) for females.
* Liver fat greater than or equal to 8% measured by MRI PDFF

Exclusion Criteria:

* Subjects with acute or chronic medical or psychiatric condition.
* Subjects with any of the following clinical laboratory abnormalities:

  * Fasting TG >400 mg/dL;
  * AST, ALT, or GGT >2.0x ULN;
  * Hemoglobin A1c (HbA1c) >7.0%;
  * Fasting plasma glucose >270 mg/dL;
  * Total bilirubin >1.5x ULN;
  * Albumin < lower limit of normal (LLN);
  * Platelet count <0.95x LLN;
  * International normalized ratio (INR) greater than or equal to 1.3.
* A positive urine test for illicit drugs.
* History of regular alcohol consumption.
* Seated systolic BP>=160 mmHg and/or diastolic BP>=100 mmHg.
* Supine 12 lead ECG demonstrating a corrected QT (QTcF) interval >450 msec or a QRS interval >120 msec.
* Subjects with an estimated GFR <60 mL/min/1.73m2.
* Evidence or diagnosis of other forms of chronic liver diseases.
* Subjects with any of the following medical conditions:

  * Any condition possibly affecting drug absorption (eg prior bariatric surgery, gastrectomy, ileal resection);
  * Diagnosis of type 1 diabetes mellitus;
  * History of congestive heart failure, unstable angina, myocardial infarction, stroke, or transient ischemic attack;
  * Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin);
  * Active placement of medical devices in/on thoracic or abdominal cavities such as pacemakers, defibrillators;
* Subjects with any anatomical or pathological abnormality that would either preclude or tend to confound the analysis of study data.
* Blood donation of approximately 1 pint or more within 60 days prior to dosing.
* Subjects taking prohibited concomitant medication(s) or those unwilling/unable to switch to permitted concomitant medication(s)
* Weight loss of greater than or equal to 5% within 1 month prior to Screening.
* Unwilling or unable to comply with the Lifestyle Requirements criteria of the protocol.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; fertile male subjects who are unwilling or unable to use highly effective method(s) of contraception.
* Investigator site staff members or Pfizer employees, including their family members, directly involved in the conduct of the study.
* Subjects with known prior treatment with or participation in a clinical trial involving any of the IPs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (29):
  - Franco Felizarta, Md, Bakersfield, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - ProSciento, Inc., Chula Vista, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Floridian Clinical Research, LLC, Hialeah, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Omega Research Maitland, Orlando, Florida
  - Accel Research Sites, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - QPS-MRA, LLC-Main Office, South Miami, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Clarity Clinical Research, East Syracuse, New York
  - High Point Clinical Trials Center, High Point, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Wake Gastroenterology, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Sterling Research Group - Mt. Auburn, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - University of Tennessee Medical Center - Radiology, Knoxville, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research-Richmond, Inc., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Calle RA, Amin NB, Carvajal-Gonzalez S, Ross TT, Bergman A, Aggarwal S, Crowley C, Rinaldi A, Mancuso J, Aggarwal N, Somayaji V, Inglot M, Tuthill TA, Kou K, Boucher M, Tesz G, Dullea R, Bence KK, Kim AM, Pfefferkorn JA, Esler WP. ACC inhibitor alone or co-administered with a DGAT2 inhibitor in patients with non-alcoholic fatty liver disease: two parallel, placebo-controlled, randomized phase 2a trials. Nat Med. 2021 Oct;27(10):1836-1848. doi: 10.1038/s41591-021-01489-1. Epub 2021 Oct 11. PMID 34635855
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3711001

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants were randomized to receive placebo (3 tablets) matched to PF-05221304 and placebo (3 tablets) matched to PF-06865571 orally, twice daily for 41 days and once on Day 42. Participants were followed up to maximum of 35 days after last dose of study drug.
- PF-05221304 15mg + Placebo: Participants were randomized to receive PF-05221304 15 milligram (mg) tablets (3 tablets, each of 5 mg) and placebo (3 tablets) matched to PF-06865571, orally, twice daily for 41 days and once on Day 42. Participants were followed up to maximum of 35 days after last dose of study drug.
- PF-06865571 300 mg + Placebo: Participants were randomized to receive PF-06865571 300 mg (3 tablets, each of 100 mg) and placebo (3 tablets) matched to PF-05221304 orally, twice daily for 41 days and once on Day 42. Participants were followed up to maximum of 35 days after last dose of study drug.
- PF-05221304 15 mg + PF-06865571 300 mg: Participants were randomized to receive PF-05221304 15 mg (3 tablets, each of 5 mg) and PF-06865571 300 mg (3 tablets, each of 100 mg) orally, twice daily for 41 days and once on Day 42. Participants were followed up to maximum of 35 days after last dose of study drug.
Period: Treatment Period (42 Days)
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Started | 14 | 29 | 28 | 28
Treated | 14 | 29 | 28 | 28
Completed | 13 | 22 | 24 | 26
Not Completed | 1 | 7 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Participants screened at other site | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 0
Not completed — Unable to attend study visits | 0 | 2 | 0 | 0
Period: Follow-Up Period (35 Days)
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Started | 13 | 22 | 24 | 26
Completed | 13 | 22 | 24 | 24
Not Completed | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of investigational product post-randomization.
Groups:
- PF-05221304 15mg + Placebo: Participants were randomized to receive PF-05221304 15 mg tablets (3 tablets, each of 5 mg) and placebo (3 tablets) matched to PF-06865571, orally, twice daily for 41 days and once on Day 42. Participants were followed up to maximum of 35 days after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg | Total
Number analyzed (Participants) | 14 | 29 | 28 | 28 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 22 | 26 | 25 | 83
  >=65 years | 4 | 7 | 2 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 15 | 10 | 46
  Male | 7 | 15 | 13 | 18 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 17 | 13 | 21 | 61
  Not Hispanic or Latino | 4 | 12 | 14 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 13 | 25 | 26 | 25 | 89
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Whole Liver Proton Density Fat Fraction (PDFF) at Day 42
Description: Magnetic resonance imaging proton density fat fraction (MRI-PDFF) technique is an established method that enables quantification of fat content in the liver. It measures the fraction of mobile protons in the liver attributable to fat content and provides whole liver coverage so that fat content can be assessed across 8 Couinaud liver segments. Whole liver PDFF = PDFFs for (Segment I + Segment II + Segment III + Segment IVa + Segment IVb + Segment V + Segment VI + Segment VII + Segment VIII) divided by total number of segments assessed.
Time Frame: Baseline, Day 42
Population: Full analysis set population included all randomized participants who received at least 1 dose of investigational product and participants were assigned to the randomized treatment regardless of what treatment was received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: percent change
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 12 | 22 | 24 | 26
percent change | 8.14 [-8.56 to 27.89] | -40.01 [-47.00 to -32.09] | -30.14 [-37.97 to -21.33] | -40.13 [-46.58 to -32.90]
Statistical Analysis 1: Comparison: Placebo vs PF-05221304 15mg + Placebo; Natural log-transformed of individual relative change from baseline to Day 42 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline whole liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale. 90% CI was calculated on difference in least square (LS) mean between groups; Test type: Superiority; p = 0.0000, ANCOVA; Difference in LS mean = -44.52, 90% CI 2-sided [-54.97 to -31.65] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 2: Comparison: Placebo vs PF-06865571 300 mg + Placebo; Natural log-transformed of individual relative change from baseline to Day 42 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline whole liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale. 90% CI was calculated on difference LS mean between groups; Test type: Superiority; p = 0.0007, ANCOVA; Difference in LS Mean = -35.40, 90% CI 2-sided [-47.40 to -20.68] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 3: Comparison: Placebo vs PF-05221304 15 mg + PF-06865571 300 mg; Natural log-transformed of individual relative change from baseline to Day 42 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline whole liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale. 90% CI was calculated on difference in LS mean between groups; Test type: Superiority; p = 0.0000, ANCOVA; Difference in LS Mean = -44.64, 90% CI 2-sided [-54.80 to -32.19] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 4: Comparison: PF-05221304 15mg + Placebo vs PF-05221304 15 mg + PF-06865571 300 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.9836, ANCOVA; Difference in LS Mean = -0.21, 90% CI 2-sided [-15.66 to 18.08] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 5: Comparison: PF-06865571 300 mg + Placebo vs PF-05221304 15 mg + PF-06865571 300 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.1233, ANCOVA; Difference in LS Mean = -14.30, 90% CI 2-sided [-27.32 to 1.06] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 6: Comparison: PF-05221304 15mg + Placebo vs PF-05221304 15 mg + PF-06865571 300 mg; Natural log-transformed of individual relative change from baseline to Day 42 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline whole liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale. 50% CI was calculated on difference in LS mean between groups; Test type: Superiority; Difference in LS Mean = -0.21, 50% CI 2-sided [-6.82 to 6.87] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model
Statistical Analysis 7: Comparison: PF-06865571 300 mg + Placebo vs PF-05221304 15 mg + PF-06865571 300 mg; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; Difference in LS Mean = -14.30, 50% CI 2-sided [-19.86 to -8.35] — LS mean difference was not a simple subtraction between LS means of groups but through statistical model

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included all serious and non-serious adverse events.
Time Frame: Baseline up to 35 days from last dose of study drug or early termination: (maximum up to Day 77)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 14 | 29 | 28 | 28
Participants
  Participants With AEs | 3 | 10 | 10 | 10
  Participants With SAEs | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Clinical chemistry: Bilirubin (milligram per deciliter [mg/dL]), direct bilirubin (mg/dL)>3.0*upper limit of normal (ULN), alanine aminotransferase international units per liter (U/L), aspartate aminotransferase (U/L), alkaline phosphatase (U/L), gamma glutamyl transferase (U/L)>5.0*ULN, urea nitrogen (mg/dL)>2.0*ULN, low density lipoprotein direct endpoint measure (mg/dL)>1.5*ULN, triglycerides (mg/dL)>2.0*ULN, creatinine based estimated glomerular filtration rate by modification of diet in renal disease equation and cystatin based eGFR by chronic kidney disease epidemiology collaboration equation (C <60 milliliter per minute per 1.73 square of meter), very low density lipoprotein (millimoles per liter), Cholesterol >2.0*ULN.
Time Frame: Baseline up to 35 days last from dose of study drug or early termination (maximum up to Day 77)
Population: Safety analysis population included all participants who received at least 1 dose of investigational product. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for laboratory abnormalities.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 14 | 29 | 27 | 26
Participants | 6 | 17 | 11 | 6

4. Secondary Outcome: Maximum Change (Increase or Decrease) From Baseline to Post-last Dose of Study Drug in Vital Signs: Blood Pressure
Description: Vital signs included systolic blood pressure, diastolic blood pressure and pulse rate.
Time Frame: Baseline, Post-last dose of study drug (up to Day 42)
Population: Safety analysis population included all participants who received at least 1 dose of investigational product post-randomization. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 14 | 29 | 28 | 26
millimeter of mercury
  Maximum increase: Systolic blood pressure | 10.8 (6.59) | 7.0 (7.77) | 9.6 (11.38) | 7.5 (12.58)
  Maximum increase: Diastolic blood pressure | 6.1 (6.86) | 3.9 (7.15) | 5.0 (7.20) | 4.3 (8.11)
  Maximum decrease: Systolic blood pressure | -9.7 (11.12) | -8.9 (7.69) | -9.2 (10.69) | -12.0 (12.54)
  Maximum decrease: Diastolic blood pressure | -6.2 (7.56) | -7.7 (7.58) | -7.3 (6.69) | -7.2 (8.09)

5. Secondary Outcome: Maximum Change (Increase or Decrease) From Baseline to Post-last Dose of Study Drug in Vital Signs: Pulse Rate
Description: Vital signs included systolic blood pressure, diastolic blood pressure and pulse rate.
Time Frame: Baseline, Post- last dose of study drug (up to Day 42)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 14 | 29 | 28 | 26
beats per minute
  Maximum increase: Pulse rate | 7.5 (8.56) | 8.1 (9.35) | 6.8 (9.13) | 6.9 (8.69)
  Maximum decrease: Pulse rate | -3.4 (7.62) | -2.9 (7.25) | -7.5 (7.47) | -5.8 (7.91)

6. Secondary Outcome: Number of Participants Meeting Pre-Specified Electrocardiogram (ECG) Criteria
Description: ECG criteria included: 1) PR interval (milliseconds [msec]): baseline greater than (>) 200 msec and maximum increase from baseline greater than or equal to (>=) 25 percent (%) or baseline less than or equal to (<=) 200 msec and maximum increase from baseline >=50%; 2) QRS interval (msec): maximum increase from baseline >=50%; 3) QT interval corrected using Fridericia's formula (QTcF): a) change from baseline >30 msec and <=60 msec, b) change from baseline >60 msec.
Time Frame: Baseline up to 35 days last dose of study drug or early termination (maximum up to Day 77)
Population: Safety analysis population included all participants who received at least 1 dose of investigational product post-randomization. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 15 mg + PF-06865571 300 mg
Number analyzed (Participants) | 14 | 29 | 28 | 26
Participants
  PR interval: %Change >=25/50%: number analyzed (Participants) | 14 | 28 | 28 | 26
  PR interval: %Change >=25/50% | 0 | 0 | 0 | 0
  QRS interval: %Change >=50% | 0 | 0 | 0 | 0
  QTcF: Change >30 msec and <=60 msec | 0 | 2 | 0 | 1
  QTcF: Change >60 msec | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days from last dose of study drug or early termination (maximum up to Day 77 days)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population included all participants who received at least 1 dose of investigational product post-randomization.
Groups:
- PF-05221304 |15mg Q12H + |PF-06865571 |300mg Q12H: Participants were randomized to receive PF-05221304 15 mg tablets and PF-06865571 300 mg tablets, orally, twice daily for 42 days. Participants were followed up to maximum of 35 days after last dose of study drug.
Arm/Group | Placebo | PF-05221304 15mg + Placebo | PF-06865571 300 mg + Placebo | PF-05221304 |15mg Q12H + |PF-06865571 |300mg Q12H
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/29 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/29 | 0/28 | 1/28
Other Adverse Events (participants affected / at risk) | 3/14 | 6/29 | 6/28 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-05221304 15mg + Placebo (N=29) | PF-06865571 300 mg + Placebo (N=28) | PF-05221304 |15mg Q12H + |PF-06865571 |300mg Q12H (N=28)
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-05221304 15mg + Placebo (N=29) | PF-06865571 300 mg + Placebo (N=28) | PF-05221304 |15mg Q12H + |PF-06865571 |300mg Q12H (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03776175/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT03776175/SAP_001.pdf